## A QUALITATIVE STUDY TO EXPLORE THE BARRIERS TO ADOPTION OF CLINICAL DECISION SUPPORT SYSTEMS (CDSS-ADOPT)

Consent Form v1.1 (06/01/2026)
NCT number pending

Medway NHS Foundation Trust Project Reference: 1366 / IRAS ID: 365984





## **Consent Form**

| Project Title | A Qualitative Study to Explore the Barriers to Adoption of Clinical Decision Support Systems |
|---|---|
| Principle investigator name | Saad Muhammad |
| IRAS Project ID | 365984 |

| | | Please |
|---|---|---|
| | | initial |
| 1. | I confirm that I have read and understood the information sheet dated// (Version) for the above study and have had the opportunity to ask questions | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my work or legal rights being affected. | |
| 3. | I understand that my responses may be looked at by responsible individuals from the research team or from regulatory authorities, or NHS Trust where it is relevant to my taking part in the research. I permit these individuals to have access to my responses. | |
| 4. | I agree to take part in the above study. | |

| Name of participant |
|---------------------|
| Date |
| Signature |





| Name of person taking consent |
|-------------------------------|
| Date |
| Signature |

Please complete in duplicate and allocate 1 form for the Participant and, 1 to be kept with filing notes (original).